CLINICAL TRIAL: NCT06256367
Title: Cariprazine Real-world Use in Bipolar I Disorder: Effectiveness, Functioning, Quality of Life, and Tolerability
Brief Title: Observational Study of Oral Cariprazine Capsules to Assess Change in Disease Activity in Adult Participants With Bipolar I Disorder
Acronym: CReW BP-I
Status: Active, not recruiting | Type: Observational
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Other Study IDs: P24-477
Record Dates: First submitted 2024-02-05; First posted 2024-02-13 (Actual); Last update posted 2025-09-23 (Actual); Status verified 2025-09

CONDITIONS: Bipolar I Disorder
Keywords: Bipolar I Disorder; Cariprazine; CReW BP-I

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Cariprazine: Participants will receive cariprazine as prescribed by their physician in routine clinical practice. The decision to initiate cariprazine should be made prior to, and independently from, the decision to participate in this study.

SUMMARY:
Bipolar I disorder (BP-I) is a common, chronic, and disabling mental illness with significant morbidity and mortality defined by episodes of mania and depression (or symptoms of both at once, known as mixed features). This prospective, observational study will examine effectiveness, functioning and quality of life outcomes in adult patients with BP-I experiencing a major depressive episode (with or without mixed features) requiring treatment and initiating treatment with cariprazine. It will examine outcomes of cariprazine treatment in a real-world setting in patients with BP-I commonly seen in clinical practices.

Cariprazine (Vraylar) is a medication indicated in the United States and Canada to treat adult patients experiencing manic, mixed or depressive episodes associated with BP-I. This study plans to enroll approximately 170 adult patients with BP-I from the United States and Canada. Cariprazine should be prescribed by the physician under the usual and customary practice of physician prescription. The decision to initiate treatment with cariprazine should be made prior to, and independently from, the patient's decision to participate in the study.

Participants will receive cariprazine as prescribed by their physician. Observational data will be collected during visits which should align to routine standard of care for a duration of up to 24 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Have a physician-confirmed diagnosis of BP-I, with or without comorbidities.
* Prescribed cariprazine as part of routine clinical practice with the intention of treating as per the approved market label, respective country indications, and by the physician under usual and customary practice of physician prescription.
* Have a Montgomery-Åsberg Depression Rating Scale (MADRS) score >= 20 at baseline.
* Have a Functioning Assessment Short Test (FAST) score >= 21 at baseline.
* Naïve to cariprazine in the current major depressive episode.

Exclusion Criteria:

* Have a medical or psychiatric condition, or planned surgical procedure, which will interfere with study participation, as judged by the investigator.
* Have a known contraindication to cariprazine including any of the following:

  * Hypersensitivity to cariprazine or any ingredient in the formulation
  * For all sites, concomitant use of strong cytochrome P450 (CYP) 3A4 inhibitors and inducers
  * For Canadian sites, as per country label, concomitant use of moderate CYP 3A4 inhibitors and inducers
* Current major depressive episode duration > 12 months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with a bipolar I disorder diagnosis experiencing a major depressive episode (with or without mixed features) requiring treatment and being prescribed cariprazine by their physician; irrespective of study participation.
Sampling Method: Probability Sample
Enrollment: 170 (Estimated)
Dates: Start 2024-04-18 (Actual); Primary Completion 2026-02 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
Change From Baseline on Montgomery-Åsberg Depression Rating Scale (MADRS) Total Score | Up to Week 12
  MADRS is a 10-item questionnaire that is rated by investigators to assess changes in depression symptoms over the past week. The individual items (apparent sadness, reported sadness, feelings of tension, reduced appetite, reduced sleep, lassitude, concentration difficulties, pessimistic thoughts, inability to feel emotions, and suicidal thoughts) are scored from 0 (no symptoms) to 6 (maximum severity) and summed for the total score (range 0 to 60). Higher scores indicate more severe depression.

SECONDARY OUTCOMES:
Change From Baseline on Functioning Assessment Short Test (FAST) Total Score | Up to Week 12
  The FAST is comprised of 24 items and assesses disability or impairment in 6 domains: autonomy, occupational functioning, financial issues, interpersonal relationships, cognitive functioning, and leisure time. FAST is administered by the investigator as an interview. Items are rated using a 4-point scale, from 0 (no difficulty) to 3 (severe difficulty) then summed for a total score. Higher scores indicate more severe impairment.

CONTACTS AND LOCATIONS:
Overall Officials: ABBVIE INC., Study Director — AbbVie
Locations (19):
- United States (11):
  - University of Alabama at Birmingham - Main /ID# 260000, Birmingham, Alabama
  - Bowman Medical Group /ID# 259989, Beverly Hills, California
  - UC Davis /ID# 259723, Sacramento, California
  - Montano Wellness LLC /ID# 259837, Cromwell, Connecticut
  - Georgia Psychiatric Consultants & Advanced Discovery Research /ID# 259975, Atlanta, Georgia
  - Omaha Insomnia and Psychiatric Services /ID# 259961, Omaha, Nebraska
  - Quest Therapeutics of Avon /ID# 259838, Avon Lake, Ohio
  - North Star Medical Research LL /ID# 259730, Middleburg Heights, Ohio
  - Rivus Wellness And Research Institute /ID# 259966, Oklahoma City, Oklahoma
  - Betts Psychiatric, PC /ID# 259737, Eugene, Oregon
  - Ut Southwestern Medical Center /Parkland Health and Hospital System /Id# 260001, Dallas, Texas
- Canada (8):
  - Chatham-Kent Clinical Trials /ID# 262414, Chatham, Ontario
  - Grand River Hospital /ID# 263962, Kitchener, Ontario
  - Sunny Johnson Medical Research Associates /ID# 267713, Mississauga, Ontario
  - Southlake Regional Health Centre /ID# 264212, Newmarket, Ontario
  - START Clinic for Mood and Anxiety Disorders /ID# 262416, Toronto, Ontario
  - Institut universitaire en santé mentale de Montréal /ID# 264665, Montreal, Quebec
  - Clinique Woodward /ID# 264050, Sherbrooke, Quebec
  - Douglas Mental Health University Institute /ID# 262048, Verdun, Quebec

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: Related Info — https://www.abbvieclinicaltrials.com/study/?id=P24-477